CLINICAL TRIAL: NCT00804167
Title: Profile of Hypertensive Patients Aged of 75 Years and Older Seen in General Practitioner According to Their Renal Damage.
Brief Title: National Survey on Hypertension
Acronym: SERENITE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2008/1
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Hypertensive patients aged of 75 years and older; renal damage; Clinical characteristics of hypertensive patients aged of 75 years and older seen in general practitioner consultation according to their renal damage
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Describe the clinical characteristics of hypertensive patients aged of 75 years and older seen in general practitioner consultation according to their renal damage

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 75 years or older
* With a diagnosis of Hypertension treated or not, seen in general practitioner consultation
* Who has given his/her consent to participate to the study.

Exclusion Criteria:

* Patient who participated to a clinical trial

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The first 3 consecutive patients seen during the GP's visit with a diagnosis of Hypertension and with renal damage
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2008-12; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Describe the clinical characteristics of hypertensive patients aged of 75 years and older seen in general practitioner consultation according to their renal damage | once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (1291):
- France (1291):
  - Research Site, Abbeville
  - Research Site, Ablon-sur-Seine
  - Research Site, Achères
  - Research Site, Achicourt
  - Research Site, Ahuy
  - Research Site, Aigre
  - Research Site, Aire-sur-la-Lys
  - Research Site, Aix-en-Provence
  - Research Site, Aixe-sur-Vienne
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Allonnes
  - Research Site, Allouagne
  - Research Site, Althen-des-Paluds
  - Research Site, Amagne
  - Research Site, Ambert
  - Research Site, Ambierle
  - Research Site, Ambleteuse
  - Research Site, Amboise
  - Research Site, Amfreville-la-Mi-Voie
  - Research Site, Amiens
  - Research Site, Amphion-les-Bains
  - Research Site, Anduze
  - Research Site, Angers
  - Research Site, Anglet
  - Research Site, Aniane
  - Research Site, Annecy
  - Research Site, Annonay
  - Research Site, Anvin
  - Research Site, Anzin
  - Research Site, Apt
  - Research Site, Arbois
  - Research Site, Arcachon
  - Research Site, Arcis-sur-Aube
  - Research Site, Ardres
  - Research Site, Arès
  - Research Site, Argeles
  - Research Site, Argentré-du-Plessis
  - Research Site, Arles
  - Research Site, Armentières
  - Research Site, Arpajon
  - Research Site, Arras
  - Research Site, Artannes-sur-Indre
  - Research Site, Arudy
  - Research Site, Asnières-sur-Seine
  - Research Site, Athies
  - Research Site, Aubenas
  - Research Site, Aubergenville
  - Research Site, Aubervilliers
  - Research Site, Auby
  - Research Site, Auch
  - Research Site, Auchy-les-Mines
  - Research Site, Auchy-lès-Hesdin
  - Research Site, Audincourt
  - Research Site, Audun-le-Roman
  - Research Site, Aulnoy-lez-Valenciennes
  - Research Site, Aulnoye-Aymeries
  - Research Site, Aumale
  - Research Site, Auneuil
  - Research Site, Aups
  - Research Site, Aurillac
  - Research Site, Authon-du-Perche
  - Research Site, Autun
  - Research Site, Auxerre
  - Research Site, Auxonne
  - Research Site, Availles-en-Châtellerault
  - Research Site, Avensan
  - Research Site, Avesnes-le-Sec
  - Research Site, Avesnes-les-Aubert
  - Research Site, Avignon
  - Research Site, Avoine
  - Research Site, Avranches
  - Research Site, Avricourt
  - Research Site, Avrillé
  - Research Site, Azerailles
  - Research Site, Bachant
  - Research Site, Badevel
  - Research Site, Bages
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baignes STE Radegonde
  - Research Site, Bailleul
  - Research Site, Bains
  - Research Site, Bais
  - Research Site, Balbigny
  - Research Site, Balma
  - Research Site, Banyuls de la Marenda
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Barjols
  - Research Site, Barlin
  - Research Site, Bassussarry
  - Research Site, Bastelicaccia
  - Research Site, Bastia
  - Research Site, Baume-les-Dames
  - Research Site, Bayonne
  - Research Site, Beaucouzé
  - Research Site, Beaulieu-sous-la-Roche
  - Research Site, Beaumont
  - Research Site, Beaumont-en-Véron
  - Research Site, Beaurepaire
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Beauzelle
  - Research Site, Behren-lès-Forbach
  - Research Site, Belfort
  - Research Site, Bellac
  - Research Site, Bellegarde-sur-Valserine
  - Research Site, Belleville-sur-Meuse
  - Research Site, Belvèze-du-Razès
  - Research Site, Belz
  - Research Site, Benfeld
  - Research Site, Berck
  - Research Site, Bergerac
  - Research Site, Bergholtz
  - Research Site, Bergues
  - Research Site, Berre-l'Étang
  - Research Site, Bersée
  - Research Site, Berson
  - Research Site, Bertrichamps
  - Research Site, Bessèges
  - Research Site, Bethoncourt
  - Research Site, Bettancourt-la-Ferrée
  - Research Site, Betton
  - Research Site, Betz
  - Research Site, Beynes
  - Research Site, Bégard
  - Research Site, Bérat
  - Research Site, Bétaille
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Bienvillers-au-Bois
  - Research Site, Bignan
  - Research Site, Blaesheim
  - Research Site, Blagnac
  - Research Site, Blamont
  - Research Site, Blanquefort
  - Research Site, Bletterans
  - Research Site, Blois
  - Research Site, Bobigny
  - Research Site, Boën-sur-Lignon
  - Research Site, Bois-Colombes
  - Research Site, Bois-le-Roi
  - Research Site, Boissy-Saint-Léger
  - Research Site, Bolbec
  - Research Site, Bondoufle
  - Research Site, Bondues
  - Research Site, Bondy
  - Research Site, Bonsecours
  - Research Site, Bornel
  - Research Site, Bosc-le-Hard
  - Research Site, Bosmie-l'Aiguille
  - Research Site, Bouafle
  - Research Site, Boucau
  - Research Site, Bouëx
  - Research Site, Bouguenais
  - Research Site, Boujan-sur-Libron
  - Research Site, Boulbon
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Gesse
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourg de Joué-sur-Erdre
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourg-lès-Valence
  - Research Site, Bousse
  - Research Site, Bracieux
  - Research Site, Braine
  - Research Site, Bram
  - Research Site, Branne
  - Research Site, Brax
  - Research Site, Bresles
  - Research Site, Bressuire
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Bretignolles-sur-Mer
  - Research Site, Bretteville-l'Orgueilleuse
  - Research Site, Brignais
  - Research Site, Bron
  - Research Site, Brouvelieures
  - Research Site, Broût-Vernet
  - Research Site, Bruay-sur-l'Escaut
  - Research Site, Bruère-Allichamps
  - Research Site, Brunoy
  - Research Site, Bry-sur-Marne
  - Research Site, Bubry
  - Research Site, Buchelay
  - Research Site, Burie
  - Research Site, Bussy-en-Othe
  - Research Site, Buxy
  - Research Site, Cabannes
  - Research Site, Cachan
  - Research Site, Caen
  - Research Site, Calais
  - Research Site, Caluire-et-Cuire
  - Research Site, Camblanes
  - Research Site, Cambrai
  - Research Site, Cambremer
  - Research Site, Camors
  - Research Site, Cancon
  - Research Site, Canet-en-Roussillon
  - Research Site, Canet-Plage
  - Research Site, Canéjan
  - Research Site, Cannes
  - Research Site, Cannes La Bocca
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Cappelle-en-Pévèle
  - Research Site, Carantec
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carhaix-Plouguer
  - Research Site, Carignan
  - Research Site, Carpentras
  - Research Site, Carpiquet
  - Research Site, Carquefou
  - Research Site, Carrières-sur-Seine
  - Research Site, Carrouges
  - Research Site, Carry-le-Rouet
  - Research Site, Carvin
  - Research Site, Cassis
  - Research Site, Castanet-Tolosan
  - Research Site, Castelnaudary
  - Research Site, Castets
  - Research Site, Castéra-Verduzan
  - Research Site, Castres
  - Research Site, Caussade
  - Research Site, Cavignac
  - Research Site, Cepoy
  - Research Site, Cerizay
  - Research Site, Cernay
  - Research Site, Cérences
  - Research Site, Chabris
  - Research Site, Chaillevette
  - Research Site, Chalais
  - Research Site, Challain-la-Potherie
  - Research Site, Challes-les-Eaux
  - Research Site, Chambéry
  - Research Site, Chambon-sur-Voueize
  - Research Site, Champagnole
  - Research Site, Champigneulles
  - Research Site, Champigné
  - Research Site, Champigny-sur-Marne
  - Research Site, Chanac
  - Research Site, Chanteheux
  - Research Site, Chantepie
  - Research Site, Chantilly
  - Research Site, Chapelle Saint Martin Plaine
  - Research Site, Charleville-Mézières
  - Research Site, Charmes
  - Research Site, Charmoy
  - Research Site, Chartres
  - Research Site, Chartres-de-Bretagne
  - Research Site, Chartrettes
  - Research Site, Charvieu-Chavagneux
  - Research Site, Chasseneuil-du-Poitou
  - Research Site, Chatou
  - Research Site, Chaumont
  - Research Site, Chaville
  - Research Site, Chazelles-sur-Lyon
  - Research Site, Châbons
  - Research Site, Châlette-sur-Loing
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-Chinon(Ville)
  - Research Site, Château-Gontier
  - Research Site, Château-Thierry
  - Research Site, Châteaumeillant
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châteauneuf-sur-Isère
  - Research Site, Châteauneuf-sur-Sarthe
  - Research Site, Châtel-Montagne
  - Research Site, Châtelaillon-Plage
  - Research Site, Châtellerault
  - Research Site, Châtenay-Malabry
  - Research Site, Châtillon-Coligny
  - Research Site, Chemellier
  - Research Site, Cheminot
  - Research Site, Chenôve
  - Research Site, Cherbourg Octeville
  - Research Site, Cherisy
  - Research Site, Cherves-Richemont
  - Research Site, Chevaigné
  - Research Site, Chevigny-Saint-Sauveur
  - Research Site, Chevry-Cossigny
  - Research Site, Chiry-Ourscamp
  - Research Site, Cholet
  - Research Site, Ciboure
  - Research Site, Cinq-Mars-la-Pile
  - Research Site, Cirey-sur-Vezouze
  - Research Site, Ciry-le-Noble
  - Research Site, Claix
  - Research Site, Clamart
  - Research Site, Clary
  - Research Site, Clermont-Ferrand
  - Research Site, Clerval
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Cluis
  - Research Site, Cognac
  - Research Site, Coignières
  - Research Site, Colmar
  - Research Site, Colombes
  - Research Site, Colombier-Fontaine
  - Research Site, Colomiers
  - Research Site, Combrit
  - Research Site, Commentry
  - Research Site, Conches-en-Ouche
  - Research Site, Conchy-les-Pots
  - Research Site, Condat-sur-Vienne
  - Research Site, Contes
  - Research Site, Corbehem
  - Research Site, Cordes-sur-Ciel
  - Research Site, Corme-Royal
  - Research Site, Corsept
  - Research Site, Corseul
  - Research Site, Cotignac
  - Research Site, Coubon
  - Research Site, Couhé
  - Research Site, Coulanges-lès-Nevers
  - Research Site, Coulonges-sur-lAutize
  - Research Site, Courbevoie
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courpière
  - Research Site, Courseulles-sur-Mer
  - Research Site, Courtalain
  - Research Site, Coussac-Bonneval
  - Research Site, Coutances
  - Research Site, Coutouvre
  - Research Site, Couzeix
  - Research Site, Coye-la-Forêt
  - Research Site, Crach
  - Research Site, Cravanche
  - Research Site, Creil
  - Research Site, Crèvecœur-le-Grand
  - Research Site, Crécy-la-Chapelle
  - Research Site, Croissy-sur-Seine
  - Research Site, Croix
  - Research Site, Cros-de-Cagnes
  - Research Site, Crosne
  - Research Site, Crozant
  - Research Site, Cubjac
  - Research Site, Cuers
  - Research Site, Cugand
  - Research Site, Cuise-la-Motte
  - Research Site, Culoz
  - Research Site, Dambach-la-Ville
  - Research Site, Davézieux
  - Research Site, Deauville
  - Research Site, Decazeville
  - Research Site, Deyvillers
  - Research Site, Décines-Charpieu
  - Research Site, Déville-lès-Rouen
  - Research Site, Dieppe
  - Research Site, Dieuze
  - Research Site, Digoin
  - Research Site, Dijon
  - Research Site, Dinard
  - Research Site, Divion
  - Research Site, Dole
  - Research Site, Domont
  - Research Site, Donnemarie-Dontilly
  - Research Site, Donville-les-Bains
  - Research Site, Dormans
  - Research Site, Douarnenez
  - Research Site, Douchy-les-Mines
  - Research Site, Doudeville
  - Research Site, Doué-la-Fontaine
  - Research Site, Douvaine
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Draveil
  - Research Site, Dunières
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Eauze
  - Research Site, Enghien-les-Bains
  - Research Site, Ermont
  - Research Site, Ernée
  - Research Site, Escaudain
  - Research Site, Esquerdes
  - Research Site, Estivareilles
  - Research Site, Estrées-Saint-Denis
  - Research Site, Eyguières
  - Research Site, Eyragues
  - Research Site, Échirolles
  - Research Site, Écouflant
  - Research Site, Écully
  - Research Site, Éguilles
  - Research Site, Éguzon-Chantôme
  - Research Site, Épernon
  - Research Site, Épierre
  - Research Site, Épinal
  - Research Site, Épinay-sur-Seine
  - Research Site, Épron
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étalondes
  - Research Site, Étretat
  - Research Site, Évaux-les-Bains
  - Research Site, Évron
  - Research Site, Ézy-sur-Eure
  - Research Site, Fabrezan
  - Research Site, Faches-Thumesnil
  - Research Site, Faramans
  - Research Site, Fayence
  - Research Site, Fegersheim
  - Research Site, Felletin
  - Research Site, Fenioux
  - Research Site, Fenouillet
  - Research Site, Ferrière-la-Grande
  - Research Site, Ferrières-en-Gâtinais
  - Research Site, Feucherolles
  - Research Site, Feuchy
  - Research Site, Feurs
  - Research Site, Fère-en-Tardenois
  - Research Site, Fécamp
  - Research Site, Firminy
  - Research Site, Fitz-James
  - Research Site, Fleury
  - Research Site, Flize
  - Research Site, Florange
  - Research Site, Florensac
  - Research Site, Fondettes
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontenay-aux-Roses
  - Research Site, Fontenilles
  - Research Site, Fontès
  - Research Site, Fontvieille
  - Research Site, Forbach
  - Research Site, Forges-les-Eaux
  - Research Site, Fort-Mardyck
  - Research Site, Fougères
  - Research Site, Fouras
  - Research Site, Fourneaux
  - Research Site, Fourques
  - Research Site, Franconville
  - Research Site, Frasne
  - Research Site, Fresnes-sur-Escaut
  - Research Site, Fréjus
  - Research Site, Froideconche
  - Research Site, Fromentine
  - Research Site, Frontenay-Rohan-Rohan
  - Research Site, Frouard
  - Research Site, Furiani
  - Research Site, Fussy
  - Research Site, Gabian
  - Research Site, Gagny
  - Research Site, Gamaches
  - Research Site, Garches
  - Research Site, Gardonne
  - Research Site, Gargenville
  - Research Site, Garges-lès-Gonesse
  - Research Site, Garons
  - Research Site, Gauriac
  - Research Site, Genlis
  - Research Site, Gennevilliers
  - Research Site, Gentilly
  - Research Site, Gerstheim
  - Research Site, Gières
  - Research Site, Giraumont
  - Research Site, Gironde-sur-Dropt
  - Research Site, Givet
  - Research Site, Glageon
  - Research Site, Golbey
  - Research Site, Gondrecourt-le-Château
  - Research Site, Gonneville-la-Mallet
  - Research Site, Gontaud-de-Nogaret
  - Research Site, Gorcy
  - Research Site, Gourdon
  - Research Site, Gournay-en-Bray
  - Research Site, Goven
  - Research Site, Granges-sur-Vologne
  - Research Site, Gratentour
  - Research Site, Graulhet
  - Research Site, Gray-la-Ville
  - Research Site, Grenoble
  - Research Site, Gréasque
  - Research Site, Griesheim-près-Molsheim
  - Research Site, Grièges
  - Research Site, Gruffy
  - Research Site, Grury
  - Research Site, Guénange
  - Research Site, Guéret
  - Research Site, Guignicourt
  - Research Site, Guipry
  - Research Site, Hagetmau
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Hanches
  - Research Site, Hangenbieten
  - Research Site, Hanvec
  - Research Site, Hardelot-Plage
  - Research Site, Harnes
  - Research Site, Hautmont
  - Research Site, Hazebrouck
  - Research Site, Hellemmes-Lille
  - Research Site, Hem
  - Research Site, Herbault
  - Research Site, Hettange-Grande
  - Research Site, Heyrieux
  - Research Site, Hostens
  - Research Site, Houdan
  - Research Site, Houilles
  - Research Site, Houlgate
  - Research Site, Hundling
  - Research Site, Hyères
  - Research Site, Illkirch-Graffenstaden
  - Research Site, Inchy
  - Research Site, Irigny
  - Research Site, Isbergues
  - Research Site, Issoudun
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivry-sur-Seine
  - Research Site, Iwuy
  - Research Site, Izeaux
  - Research Site, Janzé
  - Research Site, Jarny
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jassans-Riottier
  - Research Site, Jeumont
  - Research Site, Joncherey
  - Research Site, Jonquières
  - Research Site, Joué-lès-Tours
  - Research Site, Jouy-le-Châtel
  - Research Site, Juan-les-Pins
  - Research Site, Jugon-les-Lacs
  - Research Site, Juniville
  - Research Site, Juvigné
  - Research Site, Knutange
  - Research Site, L'Ardoise
  - Research Site, L'Escarène
  - Research Site, L'Isle-Adam
  - Research Site, La Baule-Escoublac
  - Research Site, La Bâtie-Neuve
  - Research Site, La Bouilladisse
  - Research Site, La Bourboule
  - Research Site, La Cambe
  - Research Site, La Capelle-lès-Boulogne
  - Research Site, La Celle-Saint-Cloud
  - Research Site, La Chapelle-Montligeon
  - Research Site, La Chapelle-sur-Erdre
  - Research Site, La Courneuve
  - Research Site, La Couronne
  - Research Site, La Crau
  - Research Site, La Destrousse
  - Research Site, La Ferrière
  - Research Site, La Ferrière-aux-Étangs
  - Research Site, La Ferté-Frênel
  - Research Site, La Ferté-Gaucher
  - Research Site, La Ferté-Milon
  - Research Site, La Fouillade
  - Research Site, La Garde
  - Research Site, La Garenne-Colombes
  - Research Site, La Garnache
  - Research Site, La Grand-Combe
  - Research Site, La Grande-Motte
  - Research Site, La Haye-du-Puits
  - Research Site, La Haye-Pesnel
  - Research Site, La Jubaudière
  - Research Site, La Londe
  - Research Site, La Londe-les-Maures
  - Research Site, La Madeleine
  - Research Site, La Membrolle-sur-Choisille
  - Research Site, La Mézière
  - Research Site, La Motte-Servolex
  - Research Site, La Mulatière
  - Research Site, La Réole
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochefoucauld
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Tranche-sur-Mer
  - Research Site, La Varenne-Saint-Hilaire
  - Research Site, La Walck
  - Research Site, Labastide-Murat
  - Research Site, Labastide-Saint-Georges
  - Research Site, Labergement STE Marie
  - Research Site, Lacaune
  - Research Site, Lacrouzette
  - Research Site, Lagord
  - Research Site, Lambersart
  - Research Site, Lampertheim
  - Research Site, Landerneau
  - Research Site, Landéan
  - Research Site, Lanildut
  - Research Site, Lannilis
  - Research Site, Lannion
  - Research Site, Lanouaille
  - Research Site, Lanvéoc
  - Research Site, Lanvollon
  - Research Site, Lapalisse
  - Research Site, Lapouyade
  - Research Site, Lapugnoy
  - Research Site, Larche
  - Research Site, Largentière
  - Research Site, Lassigny
  - Research Site, Latresne
  - Research Site, Laval
  - Research Site, Lavernose-Lacasse
  - Research Site, Le Blanc
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Bois-dOingt
  - Research Site, Le Bourg-d'Oisans
  - Research Site, Le Bourget-du-Lac
  - Research Site, Le Breuil-en-Auge
  - Research Site, Le Bugue
  - Research Site, Le Cannet
  - Research Site, Le Châtelet-en-Brie
  - Research Site, Le Chesne
  - Research Site, Le Clion-sur-Mer
  - Research Site, Le Donjon
  - Research Site, Le Faouët
  - Research Site, Le Havre
  - Research Site, Le Mans
  - Research Site, Le Mesnil-Esnard
  - Research Site, Le Mée-sur-Seine
  - Research Site, Le Monastier-sur-Gazeille
  - Research Site, Le Mont-Dore
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Pertre
  - Research Site, Le Péage-de-Roussillon
  - Research Site, Le Pontet
  - Research Site, Le Portel
  - Research Site, Le Pradet
  - Research Site, Le Rheu
  - Research Site, Le Rouret
  - Research Site, Le Rove
  - Research Site, Le Russey
  - Research Site, Le Soler
  - Research Site, Le Taillan-Médoc
  - Research Site, Le Touquet-Paris-Plage
  - Research Site, Le Touvet
  - Research Site, Le Tréport
  - Research Site, Le Vésinet
  - Research Site, Lectoure
  - Research Site, Lens
  - Research Site, Les Bordes-sur-Arize
  - Research Site, Les Clayes-sous-Bois
  - Research Site, LES Eyzies Tayac Sireuil
  - Research Site, Les Échelles
  - Research Site, Les Grandes-Ventes
  - Research Site, Les Lilas
  - Research Site, Les Loges
  - Research Site, Les Martres-de-Veyre
  - Research Site, Les Mureaux
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Pieux
  - Research Site, Les Ponts-de-Cé
  - Research Site, Les Sables-d'Olonne
  - Research Site, Lescar
  - Research Site, Lesconil
  - Research Site, Leyme
  - Research Site, Lezoux
  - Research Site, Lésigny
  - Research Site, Lévignac
  - Research Site, Lézignan-Corbières
  - Research Site, LIEU DIT Carnon Plage
  - Research Site, Liffol-le-Grand
  - Research Site, Lignan-sur-Orb
  - Research Site, Ligny-en-Barrois
  - Research Site, Ligugé
  - Research Site, Lille
  - Research Site, Limay
  - Research Site, Limoges
  - Research Site, Limoux
  - Research Site, Lingolsheim
  - Research Site, Loches
  - Research Site, Lombez
  - Research Site, Lomme
  - Research Site, Longué-Jumelles
  - Research Site, Loos-en-Gohelle
  - Research Site, Lorgues
  - Research Site, Lorient
  - Research Site, Louannec
  - Research Site, Loudes
  - Research Site, Loudun
  - Research Site, Loué
  - Research Site, Lourdes
  - Research Site, Lourmarin
  - Research Site, Louverné
  - Research Site, Louvigné-de-Bais
  - Research Site, Louvigné-du-Désert
  - Research Site, Loyettes
  - Research Site, Lunel
  - Research Site, Lunel-Viel
  - Research Site, Lunéville
  - Research Site, Lury-sur-Arnon
  - Research Site, Lussac-les-Châteaux
  - Research Site, Lyon
  - Research Site, L’Isle-sur-le-Doubs
  - Research Site, Mably
  - Research Site, Madonne-et-Lamerey
  - Research Site, Maignelay-Montigny
  - Research Site, Maintenon
  - Research Site, Malissard
  - Research Site, Mallemort
  - Research Site, Malo-les-Bains
  - Research Site, Mamers
  - Research Site, Manciet
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Manduel
  - Research Site, Mantes-la-Jolie
  - Research Site, Mantes-la-Ville
  - Research Site, Marange-Silvange
  - Research Site, Marcilloles
  - Research Site, Marcilly-en-Villette
  - Research Site, Marcq-en-Barœul
  - Research Site, Mareuil-sur-Lay-Dissais
  - Research Site, Marguerittes
  - Research Site, Marignane
  - Research Site, Marlenheim
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marmande
  - Research Site, Marmoutier
  - Research Site, Maromme
  - Research Site, Marquion
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseille
  - Research Site, Marspich
  - Research Site, Martignas-sur-Jalle
  - Research Site, Martigues
  - Research Site, Martin-Église
  - Research Site, Maubeuge
  - Research Site, Maubourguet
  - Research Site, Mauguio
  - Research Site, Maule
  - Research Site, Mauléon-Licharre
  - Research Site, Maurecourt
  - Research Site, Maurepas
  - Research Site, Mauriac
  - Research Site, Mauvezin
  - Research Site, Maxéville
  - Research Site, Mayenne
  - Research Site, Mazan
  - Research Site, Meaux
  - Research Site, Melun
  - Research Site, Mennecy
  - Research Site, Mensignac
  - Research Site, Menthon-Saint-Bernard
  - Research Site, Mer
  - Research Site, Merkwiller-Pechelbronn
  - Research Site, Mesvres
  - Research Site, Metz
  - Research Site, Meudon
  - Research Site, Meyrueis
  - Research Site, Meyzieu
  - Research Site, Méjannes-lès-Alès
  - Research Site, Mérignac
  - Research Site, Mézidon-Canon
  - Research Site, Mimizan
  - Research Site, Miramas
  - Research Site, Mittersheim
  - Research Site, Modane
  - Research Site, Moissac
  - Research Site, Molsheim
  - Research Site, Moncé-en-Belin
  - Research Site, Moncrabeau
  - Research Site, Mondelange
  - Research Site, Mondeville
  - Research Site, Monéteau
  - Research Site, Mons-en-Laonnois
  - Research Site, Mont-Saint-Martin
  - Research Site, Montauban
  - Research Site, Montauroux
  - Research Site, Montbard
  - Research Site, Montbrison
  - Research Site, Montdidier
  - Research Site, Montescot
  - Research Site, Montesson
  - Research Site, Monteux
  - Research Site, Montfavet
  - Research Site, Montfermeil
  - Research Site, Montgeron
  - Research Site, Montigny-le-Roi
  - Research Site, Montigny-sur-Loing
  - Research Site, Montluçon
  - Research Site, Montluel
  - Research Site, Montmagny
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montreuil-l'Argillé
  - Research Site, Montreuil-sur-Ille
  - Research Site, Montrevault
  - Research Site, Montrevel-en-Bresse
  - Research Site, Montrouge
  - Research Site, Montry
  - Research Site, Monts-sur-Guesnes
  - Research Site, Montussan
  - Research Site, Morangis
  - Research Site, Moret-sur-Loing
  - Research Site, Moreuil
  - Research Site, Morlaàs
  - Research Site, Morlaix
  - Research Site, Morsang-sur-Orge
  - Research Site, Moulay
  - Research Site, Moulins-Engilbert
  - Research Site, Mouriès
  - Research Site, Moussey
  - Research Site, Mouvaux
  - Research Site, Moÿ-de-l'Aisne
  - Research Site, Mozac
  - Research Site, Mugron
  - Research Site, Mur-de-Barrez
  - Research Site, Mussidan
  - Research Site, Mutzig
  - Research Site, Mûrs-Erigné
  - Research Site, Nailhac
  - Research Site, Nançay
  - Research Site, Nangis
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Nasbinals
  - Research Site, Naucelle
  - Research Site, Naveil
  - Research Site, Nemours
  - Research Site, Neuf-Mesnil
  - Research Site, Neufchef
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Neuilly-sur-Seine
  - Research Site, Neuville-sur-Saône
  - Research Site, Neuvillette
  - Research Site, Nevers
  - Research Site, Nérac
  - Research Site, Néré
  - Research Site, Nice
  - Research Site, Nieul
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-le-Roi
  - Research Site, Noirmoutier-en-l'Île
  - Research Site, Noisy-le-Roi
  - Research Site, Noisy-le-Sec
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Nouzonville
  - Research Site, Novalaise
  - Research Site, Noyal-Pontivy
  - Research Site, Noyen-sur-Sarthe
  - Research Site, Noyers-sur-Cher
  - Research Site, Noyon
  - Research Site, Oberhausbergen
  - Research Site, Octeville
  - Research Site, Ohlungen
  - Research Site, Oinville-sur-Montcient
  - Research Site, Oissel-sur-Seine
  - Research Site, Oisy-le-Verger
  - Research Site, Olby
  - Research Site, Onesse-Laharie
  - Research Site, Oradour-sur-Glane
  - Research Site, Orange
  - Research Site, Orléans
  - Research Site, Orliénas
  - Research Site, Orthez
  - Research Site, Orvault
  - Research Site, Ossès
  - Research Site, Oullins
  - Research Site, Oye-Plage
  - Research Site, Ozoir-la-Ferrière
  - Research Site, Pacé
  - Research Site, Pagny-sur-Moselle
  - Research Site, Panazol
  - Research Site, Pantin
  - Research Site, Paray-le-Monial
  - Research Site, Parçay-les-Pins
  - Research Site, Parempuyre
  - Research Site, Paris
  - Research Site, Parthenay
  - Research Site, Pau
  - Research Site, Pauillac
  - Research Site, Peillonnex
  - Research Site, Percy
  - Research Site, Perpignan
  - Research Site, Perreux
  - Research Site, Perrigny
  - Research Site, Petit-Couronne
  - Research Site, Petite-Synthe
  - Research Site, Peymeinade
  - Research Site, Peyrat-le-Château
  - Research Site, Peyrestortes
  - Research Site, Pégomas
  - Research Site, Phalsbourg
  - Research Site, Pibrac
  - Research Site, Piennes
  - Research Site, Pierrefitte-sur-Seine
  - Research Site, Pierrefort
  - Research Site, Pipriac
  - Research Site, Plabennec
  - Research Site, Plan-de-Cuques
  - Research Site, Plancoët
  - Research Site, Pleaux
  - Research Site, Plestin-les-Grèves
  - Research Site, Pleubian
  - Research Site, Pleumeur-Gautier
  - Research Site, Pléhédel
  - Research Site, Ploemeur
  - Research Site, Plouarzel
  - Research Site, Plouédern
  - Research Site, Plouvien
  - Research Site, Plouvorn
  - Research Site, Plouzané
  - Research Site, Plouzévédé
  - Research Site, Pluvigner
  - Research Site, Poitiers
  - Research Site, Poligny
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-de-Buis-lès-Quimerch
  - Research Site, Pont-de-l'Arche
  - Research Site, Pont-du-Château
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pontailler-sur-Saône
  - Research Site, Pontault-Combault
  - Research Site, Pontchâteau
  - Research Site, Pontivy
  - Research Site, Pornic
  - Research Site, Pornichet
  - Research Site, Port Leucate
  - Research Site, Port-La Nouvelle
  - Research Site, Pouilly-sur-Loire
  - Research Site, Poussan
  - Research Site, Prayssac
  - Research Site, Pressac
  - Research Site, Prignac-et-Marcamps
  - Research Site, Provins
  - Research Site, Puygouzon
  - Research Site, Quesnoy-sur-Deûle
  - Research Site, Quevauvillers
  - Research Site, Quévreville-la-Poterie
  - Research Site, Quiberon
  - Research Site, Quimper
  - Research Site, Rabastens-de-Bigorre
  - Research Site, Ramatuelle
  - Research Site, Rambervillers
  - Research Site, Rânes
  - Research Site, Reichshoffen
  - Research Site, Reichstett
  - Research Site, Reims
  - Research Site, Remiremont
  - Research Site, Renazé
  - Research Site, Rennes
  - Research Site, Revel
  - Research Site, Rezé
  - Research Site, Ribérac
  - Research Site, Rieumes
  - Research Site, Rieupeyroux
  - Research Site, Rive-de-Gier
  - Research Site, Rivehaute
  - Research Site, Rivière-sur-Tarn
  - Research Site, Rodez
  - Research Site, Rognac
  - Research Site, Rognes
  - Research Site, Rohrwiller
  - Research Site, Roisel
  - Research Site, Romagnat
  - Research Site, Romagné
  - Research Site, Romainville
  - Research Site, Romanswiller
  - Research Site, Rombas
  - Research Site, Romorantin-Lanthenay
  - Research Site, Roncey
  - Research Site, Ronchin
  - Research Site, Roncq
  - Research Site, Roquefort-sur-Soulzon
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Roullet-Saint-Estèphe
  - Research Site, Rouvres-en-Plaine
  - Research Site, Royan
  - Research Site, Roye
  - Research Site, Ruffec
  - Research Site, Rully
  - Research Site, Rumigny
  - Research Site, Rungis
  - Research Site, Sabres
  - Research Site, Sains-en-Amiénois
  - Research Site, Saint Maximin LA STE Baume
  - Research Site, Saint-Ambroix
  - Research Site, Saint-Amé
  - Research Site, Saint-Amour
  - Research Site, Saint-André-des-Eaux
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubin-lès-Elbeuf
  - Research Site, Saint-Aunès
  - Research Site, Saint-Avertin
  - Research Site, Saint-Barthélemy-de-Vals
  - Research Site, Saint-Barthélémy
  - Research Site, Saint-Beauzire
  - Research Site, Saint-Benoît
  - Research Site, Saint-Bonnet-sur-Gironde
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Christol-les-Alès
  - Research Site, Saint-Ciers-sur-Gironde
  - Research Site, Saint-Claude
  - Research Site, Saint-Clément
  - Research Site, Saint-Cloud
  - Research Site, Saint-Cyprien
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Cyr-sur-Mer
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-lès-Bourg
  - Research Site, Saint-Didier-en-Velay
  - Research Site, Saint-Dié
  - Research Site, Saint-Dizier
  - Research Site, Saint-Donat-sur-l'Herbasse
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Erme-Outre-et-Ramecourt
  - Research Site, Saint-Estève
  - Research Site, Saint-Etienne
  - Research Site, Saint-Etienne-de-Tulmont
  - Research Site, Saint-Émilion
  - Research Site, Saint-Étienne-du-Rouvray
  - Research Site, Saint-Félix-de-Lodez
  - Research Site, Saint-Fort-sur-Gironde
  - Research Site, Saint-Fulgent
  - Research Site, Saint-Gaudens
  - Research Site, Saint-Geniès-Bellevue
  - Research Site, Saint-Germain-les-Belles
  - Research Site, Saint-Germainmont
  - Research Site, Saint-Gratien
  - Research Site, Saint-Hilaire-de-Riez
  - Research Site, Saint-Hippolyte-du-Fort
  - Research Site, Saint-Jean-de-la-Ruelle
  - Research Site, Saint-Jean-des-Baisants
  - Research Site, Saint-Jean-en-Royans
  - Research Site, Saint-Julien-sur-Cher
  - Research Site, Saint-Just-Chaleyssin
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Just-le-Martel
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Laurent-Médoc
  - Research Site, Saint-Leu-la-Forêt
  - Research Site, Saint-Léon-sur-l'Isle
  - Research Site, Saint-Loubès
  - Research Site, Saint-Louis
  - Research Site, Saint-Lô
  - Research Site, Saint-Mamert-du-Gard
  - Research Site, Saint-Marcel-lès-Valence
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Martin-d'Uriage
  - Research Site, Saint-Martin-de-Crau
  - Research Site, Saint-Martin-de-Seignanx
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Martin-le-Beau
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-des-Lions
  - Research Site, Saint-Médard-d'Eyrans
  - Research Site, Saint-Médard-en-Jalles
  - Research Site, Saint-Nicolas-d'Aliermont
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Omer
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Paul-en-Chablais
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Paul-Trois-Châteaux
  - Research Site, Saint-Philbert-de-Bouaine
  - Research Site, Saint-Pierre-d'Albigny
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-des-Fleurs
  - Research Site, Saint-Pierre-du-Mont
  - Research Site, Saint-Pierre-en-Val
  - Research Site, Saint-Pierre-le-Moûtier
  - Research Site, Saint-Pourçain-sur-Sioule
  - Research Site, Saint-Priest
  - Research Site, Saint-Priest-Taurion
  - Research Site, Saint-Puy
  - Research Site, Saint-Quentin
  - Research Site, Saint-Quentin-la-Poterie
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Romain-de-Jalionas
  - Research Site, Saint-Saëns
  - Research Site, Saint-Saturnin-lès-Apt
  - Research Site, Saint-Sauveur
  - Research Site, Saint-Sauveur-le-Vicomte
  - Research Site, Saint-Sulpice-la-Pointe
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saint-Trivier-sur-Moignans
  - Research Site, Saint-Vaast-la-Hougue
  - Research Site, Saint-Yrieix-sur-Charente
  - Research Site, Sainte-Geneviève-des-Bois
  - Research Site, Saintes
  - Research Site, Salbris
  - Research Site, Salernes
  - Research Site, Salers
  - Research Site, Salies-de-Béarn
  - Research Site, Sallebœuf
  - Research Site, Salles
  - Research Site, Samer
  - Research Site, Sanary-sur-Mer
  - Research Site, Santec
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sars-Poteries
  - Research Site, Saulces-Monclin
  - Research Site, Saulieu
  - Research Site, Sauveterre-de-Béarn
  - Research Site, Savignac-les-Églises
  - Research Site, Savigny-sur-Orge
  - Research Site, Schiltigheim
  - Research Site, Schirrhein
  - Research Site, Schweighouse-sur-Moder
  - Research Site, Secondigny
  - Research Site, Sedan
  - Research Site, Seebach
  - Research Site, Segonzac
  - Research Site, Segré
  - Research Site, Seichamps
  - Research Site, Seloncourt
  - Research Site, Senones
  - Research Site, Septfonds
  - Research Site, Seraincourt
  - Research Site, Sermoise-sur-Loire
  - Research Site, Serrières
  - Research Site, Sers
  - Research Site, Serverette
  - Research Site, Seyssinet-Pariset
  - Research Site, Seyssins
  - Research Site, Sète
  - Research Site, Sèvres
  - Research Site, Sèvres-Anxaumont
  - Research Site, Sées
  - Research Site, Sélestat
  - Research Site, Sérifontaine
  - Research Site, Sérignan
  - Research Site, Signy-l'Abbaye
  - Research Site, Sinceny
  - Research Site, Sissonne
  - Research Site, Six-Fours-les-Plages
  - Research Site, Solre-le-Château
  - Research Site, Sorcy-Saint-Martin
  - Research Site, Sotteville-lès-Rouen
  - Research Site, Souchez
  - Research Site, Souillac
  - Research Site, Soullans
  - Research Site, Soyons
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Stains
  - Research Site, STE Austreberthe
  - Research Site, STE Bazeille
  - Research Site, STE Fereole
  - Research Site, STE FOY L Argentiere
  - Research Site, STE FOY LA Grande
  - Research Site, STE Gemmes SUR Loire
  - Research Site, STE Menehould
  - Research Site, STE MERE Eglise
  - Research Site, STE Savine
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Suresnes
  - Research Site, Susville
  - Research Site, Talant
  - Research Site, Talence
  - Research Site, Targon
  - Research Site, Tarnos
  - Research Site, Taulignan
  - Research Site, Tauves
  - Research Site, Teloché
  - Research Site, Tence
  - Research Site, Ternuay Melay Saint Hilaire
  - Research Site, Terville
  - Research Site, Teyran
  - Research Site, Téteghem
  - Research Site, Thann
  - Research Site, Thiais
  - Research Site, Thiers
  - Research Site, Thionville
  - Research Site, Thonon-les-Bains
  - Research Site, Thorigné-sur-Dué
  - Research Site, Thun-Saint-Amand
  - Research Site, Tilly-sur-Seulles
  - Research Site, Torcy
  - Research Site, Toufflers
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tournefeuille
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tours
  - Research Site, Tourtour
  - Research Site, Traînel
  - Research Site, Tresses
  - Research Site, Tréguier
  - Research Site, Trévières
  - Research Site, Troisfontaines
  - Research Site, Troissereux
  - Research Site, Tulle
  - Research Site, Uchaud
  - Research Site, Uriménil
  - Research Site, Ustaritz
  - Research Site, Vabres-l'Abbaye
  - Research Site, Vagney
  - Research Site, Val-de-Reuil
  - Research Site, Valence
  - Research Site, Valentigney
  - Research Site, Valenton
  - Research Site, Valff
  - Research Site, Vallauris
  - Research Site, Valras-Plage
  - Research Site, Valréas
  - Research Site, Varces-Allières-et-Risset
  - Research Site, Varennes-sur-Allier
  - Research Site, Varennes-Vauzelles
  - Research Site, Vaucresson
  - Research Site, Vaugneray
  - Research Site, Vaulx-en-Velin
  - Research Site, Veauche
  - Research Site, Velleron
  - Research Site, Venarey-les-Laumes
  - Research Site, Vendôme
  - Research Site, Verneuil-sur-Seine
  - Research Site, Verneuil-sur-Vienne
  - Research Site, Verquières
  - Research Site, Versailles
  - Research Site, Vert-Saint-Denis
  - Research Site, Vervins
  - Research Site, Veynes
  - Research Site, Vélines
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Véretz
  - Research Site, Vétheuil
  - Research Site, Vétraz-Monthoux
  - Research Site, Vézelise
  - Research Site, Vic-sur-Aisne
  - Research Site, Vic-sur-Seille
  - Research Site, Vigneux-sur-Seine
  - Research Site, Vihiers
  - Research Site, Village-Neuf
  - Research Site, Villaines-la-Juhel
  - Research Site, Villaines-sous-Malicorne
  - Research Site, Ville-d'Avray
  - Research Site, Villebernier
  - Research Site, Villebon-sur-Yvette
  - Research Site, Villedieu-sur-Indre
  - Research Site, Villefranche-de-Lauragais
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
  - Research Site, Villemeux-sur-Eure
  - Research Site, Villemoisson-sur-Orge
  - Research Site, Villemomble
  - Research Site, Villenave-d'Ornon
  - Research Site, Villeneuve-d'Ascq
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villeneuve-Tolosane
  - Research Site, Villepreux
  - Research Site, Villers-Bocage
  - Research Site, Villers-Bretonneux
  - Research Site, Villers-Cotterêts
  - Research Site, Villerupt
  - Research Site, Villette-d'Anthon
  - Research Site, Villeurbanne
  - Research Site, Villiers-sur-Loir
  - Research Site, Villiers-sur-Marne
  - Research Site, Vinay
  - Research Site, Vincennes
  - Research Site, Vineuil
  - Research Site, Violaines
  - Research Site, Vitré
  - Research Site, Vitrolles
  - Research Site, Vitry-en-Artois
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittel
  - Research Site, Vivier-au-Court
  - Research Site, Voinémont
  - Research Site, Voiron
  - Research Site, Vonnas
  - Research Site, Vrigne-aux-Bois
  - Research Site, Vue
  - Research Site, Vœuil-et-Giget
  - Research Site, Wallers
  - Research Site, Wallon-Cappel
  - Research Site, Warloy-Baillon
  - Research Site, Warmeriville
  - Research Site, Wasquehal
  - Research Site, Wattrelos
  - Research Site, Weitbruch
  - Research Site, Westhoffen
  - Research Site, Wignehies
  - Research Site, Wingersheim
  - Research Site, Wittisheim
  - Research Site, Ydes
  - Research Site, Yutz
  - Research Site, Yvré-l'Évêque
  - Research Site, Zillisheim